CLINICAL TRIAL: NCT02633059
Title: Phase 1 / 2 Trial of Idasanutlin in Combination With Ixazomib and Dexamethasone in Patients With 17p Deleted, Relapsed Multiple Myeloma
Brief Title: Idasanutlin, Ixazomib Citrate, and Dexamethasone in Treating Patients With Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MC1582; NCI-2015-02155 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NP29909 (Other: Genentech); X16066 (Other: Millennium Pharmaceuticals, Inc.); MMRC-061 (Other: MMRF); 15-003348 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Results first posted 2022-12-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Loss of Chromosome 17p; Recurrent Plasma Cell Myeloma
MeSH Terms: conditions — Chromosome 17 deletion; Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; RG7388; ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ixazomib citrate, idasanutlin, dexamethasone) (Experimental): Patients receive ixazomib citrate PO on days 1, 8, and 15 and idasanutlin PO QD on days 1-5 every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive dexamethasone PO on days 1, 8, 15, and 22 every 28 days for 12 courses at the discretion of the treating physician.
  Interventions: Drug: Dexamethasone; Drug: Idasanutlin; Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Idasanutlin — Given PO
  Other Names: RG-7388; RG7388; RO-5503781; RO5503781
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of idasanutlin and ixazomib citrate when given together with dexamethasone in treating patients with multiple myeloma that has returned after a period of improvement. Drugs used in chemotherapy, such as idasanutlin and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Ixazomib citrate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving idasanutlin, ixazomib citrate, and dexamethasone together may work better in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated doses (MTD) of idasanutlin and ixazomib (ixazomib citrate) to be used in combination with dexamethasone in patients with relapsed or refractory multiple myeloma with TP53 (17p) deletion. (Phase I) II. To evaluate the confirmed response rate of ixazomib and idasanutlin used in combination with dexamethasone in patients with relapsed or refractory multiple myeloma with TP53 (17p) deletion. (Phase II)

SECONDARY OBJECTIVES:

I. To describe the toxicities and the confirmed response rate associated with the combination of idasanutlin, ixazomib and dexamethasone. (Phase I) II. To describe the toxicities associated with the combination of idasanutlin, ixazomib and dexamethasone. (Phase II) III. To describe the complete response (CR) and very good partial response (VGPR) rates. (Phase II) IV. To assess progression-free and overall survival. (Phase II)

TERTIARY OBJECTIVES:

I. Assess murine double minute 2 (MDM2) inhibition in bone marrow plasma cells. II. Identify potential biomarkers associated with response. III. To explore the pharmacodynamic effects of idasanutlin.

OUTLINE: This is a phase I, dose-escalation study of idasanutlin and ixazomib citrate followed by a phase II study.

Patients receive ixazomib citrate orally (PO) on days 1, 8, and 15 and idasanutlin PO once daily (QD) on days 1-5 every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive dexamethasone PO on days 1, 8, 15, and 22 every 28 days for 12 courses at the discretion of the treating physician.

After completion of study treatment, patients are followed up for 30 days, every 3 months, and then every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma (MM) with deletion 17p (del17p) or monosomy 17 by fluorescence in situ hybridization (FISH) who have received at least one line of therapy
* Calculated creatinine clearance (using Cockcroft-Gault equation) >= 30 mL/min
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x the upper limit of the normal range (ULN)
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 75,000/mm^3
* Hemoglobin >= 8.0 g/dL
* NOTE: white blood count and platelet count criteria must be met without any transfusion or growth factor support
* Patients with measurable disease defined as at least one of the following:

  * Serum monoclonal protein >= 1.0 g/dL by protein electrophoresis
  * > 200 mg of monoclonal protein in the urine on 24-hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willing to follow strict birth control measures as suggested below

  * Female patients: if they are of childbearing potential (except if postmenopausal for at least 1 year before the screening visit, OR are surgically sterile), agree to one of the following:

    * Practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
  * Male patients: even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

    * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Willing to provide bone marrow and blood samples for correlative research purposes

Exclusion Criteria:

* Other malignancy requiring active therapy

  * EXCEPTIONS: Non-melanoma skin cancer, ductal carcinoma in situ (DCIS) or carcinoma-in-situ of the cervix
  * NOTE: if there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* Other co-morbidity which would interfere with patient's ability to participate in trial, e.g. uncontrolled infection, uncompensated heart or lung disease
* Other concurrent chemotherapy, radiotherapy, or any ancillary therapy considered investigational

  * NOTE: bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Patient has >= grade 2 peripheral neuropathy, or grade 1 with pain on clinical examination during the screening period
* Major surgery =< 14 days before study registration
* All CYP2C8 inhibitors, inducers, and substrates should be discontinued >= 7 days prior to registration; systemic treatment with CYP2C8 inhibitors (anastrozole, montelukast, quercetin, trimethoprim, gemfibrozil, rosiglitazone, pioglitazone), inducers (carbamazepine, phenytoin, rifabutin, rifampin), or substrates (amiodarone, repaglinide, rosiglitazone, sorafenib, torsemide) should be discontinued >= 7 days prior to registration
* Systemic treatment with strong inhibitors of CYP3A4 (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A4 inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital, Gingko biloba, St. John's wort) are not allowed =< 14 days before registration
* Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure, angina, or myocardial infarction within the past 6 months; Note: prior to study entry, any electrocardiogram (ECG) abnormality at screening must be documented by the investigator as not medically relevant
* Corrected QT (QTc) > 470 milliseconds (msec) on a 12-lead ECG obtained during the Screening period

  * Note: If a machine reading is above this value, the ECG should be reviewed by a qualified reader and confirmed on a subsequent ECG
* Known human immunodeficiency virus (HIV) positive
* Known hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergy to any of the study medications, their analogues or excipients in the various formulations
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib or idasanutlin including difficulty swallowing
* Diarrhea > grade 1, based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grading, or currently taking antidiarrheals
* Need for ongoing therapeutic anticoagulation
* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Patients that have previously been treated with ixazomib, or who participated in a blinded study with ixazomib (whether treated with ixazomib or not)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-12-30 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, M.D., Principal Investigator — Mayo Clinic
Locations (8):
- United States (8):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Dose Level 0: Phase 1: Ixazomib 4.0 mg, Idasanutlin 100 mg, and Dexamethasone 40 mg
- Phase 1: Dose Level 1: Phase 1: Ixazomib 4.0 mg, Idasanutlin 200 mg, and Dexamethasone 40 mg
- Phase 1: Dose Level 2: Phase 1: Ixazomib 4.0 mg, Idasanutlin 250 mg, and Dexamethasone 40 mg
- Phase 2: Dose Level 1: Phase 2: Ixazomib 4.0 mg, Idasanutlin 200 mg, and Dexamethasone 40 mg
Period: Overall Study
Arm/Group | Phase 1: Dose Level 0 | Phase 1: Dose Level 1 | Phase 1: Dose Level 2 | Phase 2: Dose Level 1
Started | 4 | 7 | 4 | 18
Completed | 4 | 6 | 4 | 16
Not Completed | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Dose Level 0 | Phase 1: Dose Level 1 | Phase 1: Dose Level 2 | Phase 2: Dose Level 1 | Total
Number analyzed (Participants) | 4 | 7 | 4 | 18 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (6.60) | 60.9 (8.69) | 63.0 (12.03) | 65.0 (7.65) | 64.2 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 5 | 8
  Male | 3 | 6 | 3 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 4 | 7 | 4 | 16 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2 | 4
  White | 3 | 5 | 4 | 15 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
ECOG Performance Status (PS) [Count of Participants; unit: Participants] — ECOG = 0: Fully active, able to carry on all pre-disease performance without restriction.> ECOG = 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.> ECOG = 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.> ECOG = 0 is better. ECOG = 2 is worse.
  Participants
    0 | 1 | 2 | 2 | 6 | 11
    1 | 3 | 4 | 2 | 10 | 19
    2 | 0 | 1 | 0 | 2 | 3
Mayo Clinic Stratification for Myeloma and Risk-Adapted Therapy (mSMART) [Count of Participants; unit: Participants] — Standard Risk: All others including: Trisomies t(11;14)d t(6;14).> High Risk: t(4;14) t(14;16) t(14;20) Del 17p 53 mutation Gain 1q RISS Stage 3 High Plasma Cell S-phasec GEP: High risk signature.> Standard Risk is best, High Risk is worst.
  Participants
    High Risk | 4 | 6 | 4 | 14 | 28
    Standard Risk | 0 | 1 | 0 | 4 | 5
What was the International Staging System myeloma stage? [Count of Participants; unit: Participants] — Stage I: Sβ2M < 3.5 mg/L; serum albumin ≥ 3.5 g/dL> Stage II: Sβ2M < 3.5 mg/L; serum albumin < 3.5 g/dL; or β2M 3.5 to 5.5 mg/L, irrespective of serum albumin> Stage III: Sβ2M > 5.5 mg/L> Stage I is best, Stage III is worst.
  Participants
    Stage I | 2 | 3 | 3 | 7 | 15
    Stage II | 0 | 2 | 1 | 5 | 8
    Stage III | 2 | 1 | 0 | 2 | 5
    Unknown | 0 | 0 | 0 | 4 | 4
    Missing | 0 | 1 | 0 | 0 | 1
Revised International Staging System [Count of Participants; unit: Participants] — Stage I: Sβ2M < 3.5 mg/l, Serum albumin ≥ 3.5 g/dl, Standard-risk chromosomal abnormalities (CA) by iFISH, Normal LDH> Stage II: Not R-ISS stage I or III> Stage III: Sβ2M ≥ 5.5 mg/L and either, High-risk CA by FISH> OR, High LDH> Stage I is best, Stage III is worst
  Participants
    I | 0 | 1 | 0 | 2 | 3
    II | 2 | 5 | 4 | 14 | 25
    III | 2 | 1 | 0 | 2 | 5
Serum Creatinine (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 0.8 (0.24) | 1.1 (0.60) | 0.9 (0.19) | 1.2 (0.53) | 1.1 (0.49)
Serum LDH (U/L) [Mean (Standard Deviation); unit: (U/L)] | 201.3 (43.94) | 198.7 (162.89) | 349.0 (239.56) | 259.6 (119.45) | 249.5 (144.49)
Parameter for response [Count of Participants; unit: Participants]
  Serum M-spike >= 1 g/dL and urine M-spike >= 200 mg/24 hours | 1 | 2 | 0 | 2 | 5
  Serum M-spike >= 1 g/dL only | 3 | 2 | 2 | 4 | 11
  Urine M-spike >= 200 mg/24 hours only | 0 | 0 | 0 | 8 | 8
  Serum immunoglobulin free light chain >= 10 mg/dL | 0 | 3 | 2 | 4 | 9
(If serum M-spike), parameter followed for serum M-spike [Count of Participants; unit: Participants]
  SPEP measurement | 4 | 4 | 2 | 6 | 16
  Missing | 0 | 3 | 2 | 12 | 17
Disease category [Count of Participants; unit: Participants]
  Relapsed | 4 | 4 | 1 | 15 | 24
  Refractory | 0 | 3 | 3 | 3 | 9
Prior transplant related to this cancer [Count of Participants; unit: Participants]
  Yes | 3 | 6 | 3 | 14 | 26
  No | 1 | 1 | 1 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Experienced Dose Limiting Toxicities. Maximum Tolerated Dose (MTD) of Ixazomib Citrate and Idasanutlin in Combination With Dexamethasone (Phase I)
Description: Defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients (at least 2 of a maximum of 6 new patients). DLT is graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Dose Level 0 | Phase 1: Dose Level 1 | Phase 1: Dose Level 2 | Phase 2: Dose Level 1
Number analyzed (Participants) | 4 | 7 | 4 | 18
Participants | 0 | 0 | 2 | 1

2. Primary Outcome: Rate of Confirmed Response, Defined as a Patient Who Has Achieved a Stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), or Partial Response (PR) on Two Consecutive Evaluations (Phase II)
Description: Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success proportion will be calculated.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Phase II and MTD: 6 MTD and 16 phase II accruals
Arm/Group | Phase II and MTD
Number analyzed (Participants) | 22
Participants
  PR | 2
  SD | 6
  NA | 14
  CR | 0
  VGPR | 0
  sCR | 0

3. Secondary Outcome: Incidence of Adverse Events Graded According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 (Phase I)
Description: Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Time Frame: 30 days after the last dose of study treatment, up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Dose Level 0 | Phase 1: Dose Level 1 | Phase 1: Dose Level 2
Number analyzed (Participants) | 4 | 7 | 4
Participants
  Grade 3+ Adverse Events, Regardless of Attribution | 3 | 4 | 3
  Grade 3+ Adverse Events, At Least Possibly Related | 2 | 4 | 3
  Grade 4+ Adverse Events, Regardless of Attribution | 0 | 1 | 3
  Grade 4+ Adverse Events, At Least Possibly Related | 0 | 1 | 2
  Grade 5 Adverse Events, Regardless of Attribution | 0 | 0 | 0
  Grade 5 Adverse Events, At Least Possibly Related | 0 | 0 | 0
  Grade 3+ Heme Adverse Events, Regardless of Attribution | 3 | 4 | 3
  Grade 3+ Heme Adverse Events, At Least Possibly Related | 2 | 4 | 3
  Grade 4+ Heme Adverse Events, Regardless of Attribution | 0 | 1 | 3
  Grade 4+ Heme Adverse Events, At Least Possibly Related | 0 | 1 | 2
  Grade 5 Heme Adverse Events, Regardless of Attribution | 0 | 0 | 0
  Grade 5 Heme Adverse Events, At Least Possibly Related | 0 | 0 | 0
  Grade 3+ Non-heme Adverse Events, Regardless of Attribution | 1 | 2 | 0
  Grade 3+ Non-heme Adverse Events, At Least Possibly Related | 1 | 1 | 0
  Grade 4+ Non-heme Adverse Events, Regardless of Attribution | 0 | 0 | 0
  Grade 4+ Non-heme Adverse Events, At Least Possibly Related | 0 | 0 | 0
  Grade 5 Non-heme Adverse Events, Regardless of Attribution | 0 | 0 | 0
  Grade 5 Non-heme Adverse Events, At Least Possibly Related | 0 | 0 | 0

4. Secondary Outcome: Incidence of Adverse Events Graded According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 (Phase II)
Description: The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.
Time Frame: Up to 6 months
Population: Participants who had adverse events fitting the criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Dose Level 1
Number analyzed (Participants) | 17
Participants
  Grade 3+ Adverse Events, Regardless of Attribution | 14
  Grade 3+ Adverse Events, At Least Possibly Related | 13
  Grade 4+ Adverse Events, Regardless of Attribution | 10
  Grade 4+ Adverse Events, At Least Possibly Related | 9
  Grade 5 Adverse Events, Regardless of Attribution | 2
  Grade 5 Adverse Events, At Least Possibly Related | 0
  Grade 3+ Heme Adverse Events, Regardless of Attribution | 13
  Grade 3+ Heme Adverse Events, At Least Possibly Related | 13
  Grade 4+ Heme Adverse Events, Regardless of Attribution | 9
  Grade 4+ Heme Adverse Events, At Least Possibly Related | 9
  Grade 5 Heme Adverse Events, Regardless of Attribution | 0
  Grade 5 Heme Adverse Events, At Least Possibly Related | 0
  Grade 3+ Non-heme Adverse Events, Regardless of Attribution | 5
  Grade 3+ Non-heme Adverse Events, At Least Possibly Related | 3
  Grade 4+ Non-heme Adverse Events, Regardless of Attribution | 4
  Grade 4+ Non-heme Adverse Events, At Least Possibly Related | 2
  Grade 5 Non-heme Adverse Events, Regardless of Attribution | 2
  Grade 5 Non-heme Adverse Events, At Least Possibly Related | 0

5. Secondary Outcome: Overall Survival (Phase II)
Description: The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II and MTD
Number analyzed (Participants) | 22
months | 21.0 [10.4 to NA] — Upper limit not reached due to insufficient number of participants with events

6. Secondary Outcome: Progression Free Survival (Phase II)
Description: The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II and MTD
Number analyzed (Participants) | 22
months | 3.8 [2.2 to 7.4]

7. Secondary Outcome: Rate of Complete Response (CR) (Phase II)
Description: The rate of CR will be estimated by the number of patients with a sCR or CR or divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success proportions will be calculated.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II and MTD
Number analyzed (Participants) | 22
Participants | 0

8. Secondary Outcome: Rate of Partial Response (PR) (Phase II)
Description: The rate of PR will be estimated by the number of patients with a VGPR or PR divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success proportions will be calculated.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II and MTD
Number analyzed (Participants) | 22
Participants | 2

9. Other Pre Specified Outcome: Changes in Macrophage Inhibitory Cytokine-1 (MIC) Levels
Description: Effect of inhibition of mdm2 will be assessed by measuring MIC levels. MIC levels at each time point and changes after treatment will be both graphically and quantitatively summarized and explored. Changes from baseline will be evaluated using Wilcoxon's signed rank test.
Time Frame: Baseline up to 6 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Impact of MDM2 Inhibition on Activation of p53 and Clonal Selection
Description: Impact of MDM2 inhibition on activation of p53 and clonal selection examined using gene expression profiling and exome sequencing
Time Frame: Up to 6 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Potential Biomarkers Associated With Response Determined Using Gene Expression Profiling
Description: Potential biomarkers associated with response will be assessed in an exploratory manner. Potential markers will be determined using gene expression profiling. The correlation between potential biomarkers and response (responders vs. non-responders) will be evaluated using Fisher's exact and Wilcoxon rank sum tests, where appropriate.
Time Frame: Up to 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Phase 1: Dose Level 0 | Phase 1: Dose Level 1 | Phase 1: Dose Level 2 | Phase 2: Dose Level 1
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7 | 0/4 | 2/17
Serious Adverse Events (participants affected / at risk) | 0/4 | 3/7 | 0/4 | 6/17
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7 | 4/4 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Dose Level 0 (N=4) | Phase 1: Dose Level 1 (N=7) | Phase 1: Dose Level 2 (N=4) | Phase 2: Dose Level 1 (N=17)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Dose Level 0 (N=4) | Phase 1: Dose Level 1 (N=7) | Phase 1: Dose Level 2 (N=4) | Phase 2: Dose Level 1 (N=17)
Anemia (Blood and lymphatic system disorders) | 4 (10) | 7 (26) | 4 (10) | 14 (58)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (7) | 1 (1) | 6 (18)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (9) | 3 (6) | 8 (15)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (6) | 4 (5) | 10 (21)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4) | 6 (8)
Edema limbs (General disorders) | 0 (0) | 1 (6) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 6 (15) | 3 (5) | 10 (50)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Creatinine increased (Investigations) | 0 (0) | 5 (12) | 1 (1) | 4 (16)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 3 (5)
Neutrophil count decreased (Investigations) | 3 (9) | 5 (8) | 3 (6) | 9 (19)
Platelet count decreased (Investigations) | 4 (14) | 6 (22) | 4 (10) | 15 (59)
White blood cell decreased (Investigations) | 3 (10) | 5 (13) | 3 (6) | 12 (24)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (6) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (7) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 5 (17) | 2 (3) | 8 (51)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT02633059/Prot_SAP_000.pdf